CLINICAL TRIAL: NCT06694402
Title: The Effects of Focal Muscle Vibration Combined With Exercise on Sensorimotor Activity in Individuals With Chronic Subacromial Impingement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU113082AF
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Focal Vibration; Electroencephalography; Transcranial Magnetic Stimulation; Somatosensory Dysfunction; Corticomotor Excitability; Intracortical Inhibition; Chronic Subacromial Impingement Syndrome; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Exercise Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- focal muscle vibration combined with exercise (Experimental)
  Interventions: Device: focal muscle vibration combined with exercise
- exercise alone (Active Comparator)
  Interventions: Other: exercise

INTERVENTIONS:
Device: focal muscle vibration combined with exercise — The treatment group will receive a 30-minute intervention in each session. Focal muscle vibration will be applied to the anterior and lateral parts of shoulder to give a sensory stimulation while participants are doing eaercise.
  Arms: focal muscle vibration combined with exercise
Other: exercise — The control group will receive 30-minute exercise without focal muslce vibration.
  Arms: exercise alone

SUMMARY:
Background: Subacromial impingement syndrome (SIS) is a common shoulder disorder characterized by pain, altered movement patterns, and functional impairment. Forty-four to sixty-five percents of the patients with SIS would develop chronic symptoms. Chronic subacromial impingement syndrome (CSIS) is involved in the alteration of central nervous system, such as somatosensory dysfunction and corticomotor changes. The treatments for these patients usually focus on shoulder control and strengthening exercise but no treatment has been found to be targeted on the alterations in somatosensory dysfunction. Focal muscle vibration (FMV) is a useful tool to provide proprioceptive stimulation and has showed short-term effects of improving sensorimotor performance in both healthy and diseased individuals when combined with exercise. To our knowledge, no study has used FMV combined with shoulder exercise for individuals with shoulder problems.

Purpose: To investigate the effects of FMV combined with exercise on somatosensory activity, corticomotor excitability, pain and function in individuals with CSIS.

Methods: This is a randomized control trial. We will recruit ninety subjects with CSIS to receive a 12-session treatment protocol of FMV combined with shoulder exercises. The subjects will be randomized into a treatment group or control group. While the treatment group will receive 20-minute FMV when doing strength training, the control group will have the vibrators attached on but without being turned on during strength training. Both groups will have a 10-20 minutes of shoulder control training following the FMV protocol. The outcomes will be measured before and after the 12-session treatment protocol and include measures of somatosensory activity (using Electroencephalography, EEG), corticomotor excitability (using transcranial magnetic stimulation, TMS), pressure pain threshold, depression scale, pain intensity in a numerical rating scale, and shoulder function. The somatosensory measures include somatosensory-evoked potentials and event-related potentials during arm elevation. Corticomotor measures include motor evoked potentials, active and rest motor threshold and cortical silent period as well as intracortical inhibitory and facilitatory mechanisms. Shoulder function will be measured with the disabilities of the arm, shoulder and hand scale, the patient-specific functional scale, and the global rating of change scale.

Statistical analysis: The continuous and categorical variables of basic data will be analyzed by and independent t test and a Chi-square test, respectively. A two-way mixed ANOVA will be used to test between-group and within-group intervention effects. If there is a significant interaction effect, post hoc pairwise comparisons with Bonferroni correction will be used. The alpha level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior or lateral shoulder pain ≥ 3 months
2. 18 to 65 years old
3. The most pain intensity ≥ 3/10 Pain-Numeric Scale (NRS)
4. SIS, at least 3 positive findings of the following tests:

(1) Neer's test (2) Hawkins-Kennedy test (3) Empty can test (4) Resisted external rotation test (5) Presenting painful arc during arm elevation (6) Tenderness of the rotator cuff tendons

Exclusion Criteria:

1. History of dislocation, fracture, adhesive capsulitis or surgery of upper extremity
2. Neck pain
3. Shoulder flexion or abduction less than 150 degrees
4. History of direct contact injury to the neck or upper extremities within the past 12 months
5. Brain injury and neurological impairment
6. Inflammatory cause of the pain (e.g., rheumatoid arthritis)
7. Psychosis and symptom of headache or dizziness
8. Taking centrally acting medication
9. Contraindications to the use of transcranial magnetic stimulation (TMS)
10. Received shoulder-related physical therapy or corticosteroid injections in the past three months.
11. Received high-concentration platelet-rich plasma (PRP) injections in the shoulder joint in the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Somatosensory cortical activity - Somatosensory evoked potentials | Change from baseline SEP at the completion of 12-session intervention, an average of 6 weeks
  Somatosensory evoked potentials (SEP) will be described with microvolt (µV) and millisecond (ms).
Corticomotor excitability measures - Active motor threshold | Change from baseline AMT at the completion of 12-session intervention, an average of 6 weeks
  Active motor threshold (AMT) will be described with the percentage (%) of maximum stimulator output (MSO).
Corticomotor excitability measures - Motor evoked potential | Change from baseline MEP at the completion of 12-session intervention, an average of 6 weeks
  Motor evoked potential (MEP) will be described with millivolt (mV).
Corticomotor excitability measures - Cortical silent period | Change from baseline CSP at the completion of 12-session intervention, an average of 6 weeks
  Cortical silent period (CSP) will be measured with millisecond (ms)
Corticomotor excitability measures - Short interval cortical inhibition | Change from baseline SICI at the completion of 12-session intervention, an average of 6 weeks
  Short interval cortical inhibition (SICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms
Corticomotor excitability measures - Short interval cortical facilitation | Change from baseline SICF at the completion of 12-session intervention, an average of 6 weeks
  Short interval cortical facilitation (SICF) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is above 5 ms
Corticomotor excitability measures - Interval cortical facilitation | Change from baseline ICF at the completion of 12-session intervention, an average of 6 weeks
  Interval cortical facilitation (ICF) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is above 5 ms
Corticomotor excitability measures - Long-interval intracortical inhibition | Change from baseline LICI at the completion of 12-session intervention, an average of 6 weeks
  Long-interval intracortical inhibition (LICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms

SECONDARY OUTCOMES:
Shoulder pain and function-Taiwan version of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Change from baseline DASH scores at the completion of 12-session intervention, an average of 6 weeks
  Subjects will be asked 30 items related to shoulder functional movement. The overall score ranges from 0 (no disability) to 100 (most severe disability).
Visual analogue scale (VAS) of shoulder pain | Change from baseline VAS scores at the completion of 12-session intervention, an average of 6 weeks
  Shoulder pain and instability will be measured by visual analogue scale (VAS). Subjects need to mark the point that they feel represent their perception of their current state on a 10-cm line. Scores range from 0 (no symptom) to 100 (maximum symptom).
Depression- Taiwan version of the Center for Epidemiologic Studies Depression Scale (CES-D) | Change from baseline CES-D scores at the completion of 12-session intervention, an average of 6 weeks
  Subjects will be asked 20 items to rate how often over the past week they experienced symptoms associated with depression. Response options range from 0 to 3 for each item. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Pressure pain thresholds | Change from baseline PPT at the completion of 12-session intervention, an average of 6 weeks
  Pressure pain threshold (PPT) of bilateral upper trapezius, levator scapulae, infraspinatus, pectoralis major, biceps brachii, middle deltoid and tibialis anterior will each be averaged and will be described with kg/cm2.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chaio Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan